CLINICAL TRIAL: NCT01320137
Title: A Study in Adult Subjects With Allergy to Support the Development of Immunological Assays
Brief Title: Study in Allergic Adults to Support the Development of Immunological Assays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 115315
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Immunologic Tests
Keywords: Immunological assay; Birch allergy

ARMS (2):
- Allergy Group (Other): Subjects with ages ranging from 18-45 years and inclusive, presenting symptomatic allergy to birch pollen.
  Interventions: Procedure: Blood withdrawal
- Control Group (Other): Subjects with ages ranging from 18-45 years and inclusive, with no known allergies.
  Interventions: Procedure: Blood withdrawal

INTERVENTIONS:
Procedure: Blood withdrawal — Blood sampling

SUMMARY:
The purpose of this study is to develop and characterize immunological assays on blood samples.

DETAILED DESCRIPTION:
This is a clinical study in which there is no vaccine administered. It is designed for research purposes such as developing immunological assays.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Healthy subjects (except the condition studied in the ALLERGY group).
* A male or female between, and including 18 and 45 years of age at the time of study start.
* Subject presenting moderate to severe clinical symptoms of allergy within the week before enrolment (only for ALLERGY group).
* Subjects suffering from seasonal allergy to birch pollen previously documented by a medical history (only for ALLERGY group).
* A positive skin prick test response realised and/or a positive test for specific IgE against birch within the last 5 years (only for ALLERGY group).

Exclusion Criteria:

* Any known or clinical signs of anaemia or any condition that would preclude the drawing of blood as described in the protocol.
* Receipt of blood products 120 days prior to study visit.
* Receipt of immunoglobulin 120 days prior to study visit.
* Use of any investigational or non-registered product within 30 days preceding the study visit.
* Concurrently participating in another clinical study, at the time of the study visit, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history.
* Any confirmed or suspected autoimmune or inflammatory disorders.
* Administration of systemic or inhaled anti-inflammatory medications and, in particular, inhaled corticoid-steroids and cromoglycates within 30 days preceding the study visit. Purely local medications such as intranasal steroids or systemic symptomatic medications such as antihistamines and beta agonists are allowed.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the study visit.
* Pregnant or lactating female.
* Any past or current birch-specific immunotherapy (only for ALLERGY group).
* Any allergic disease as established by medical history before study start (only for CONTROL group).
* Family history of allergic diseases in the first degree family members (only for CONTROL group).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-03-31 (Actual); Primary Completion 2011-05-11 (Actual); Study Completion 2011-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Belgium (2):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, La Louvière

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allergy Group | Control Group
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allergy Group | Control Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.1 (7.44) | 28.6 (6.92) | 29.35 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 19 | 45
  Male | 14 | 21 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Subject Responders With Antigen Specific Lymphocytes T Helper 2 (Th2) Cluster of Differentiation 4+ (CD4+) T Cells Expressing Cytokines
Description: Among cytokines expressed were interleukin-4 (IL-4), interleukin-5 (IL-5) and/or interleukin-13 (IL-13), as measured by flow cytometry and multiplex assays.
  Responders were defined as subjects with a concentration after Bet v 1 stimulation above Percentile 95 (P95) (determined on Betula verucossa 1[Bet v 1] Bromodeoxyuridine + [BrdU+] subjects) of all concentrations after medium only stimulation
Time Frame: At Day 0
Population: The According-To-Protocol (ATP) cohort, Bet v 1 BrdU+ subjects included all subjects from the ATP cohort for which proliferation of peripheral blood mononuclear cells (PBMCs) with the birch pollen allergen Bet v 1 was observed after 96 hours.
Measure: Number; unit: Subjects
Arm/Group | Allergy Group | Control Group
Number analyzed (Participants) | 10 | 3
Subjects
  IL-13 | 7 | 1
  IL-5 | 7 | 0

2. Primary Outcome: Number of Subject Responders With Antigen Specific Th2 CD4+ T Cells Expressing Cytokines - Amended Definition
Description: Among cytokines expressed were IL-4, IL-5 and/or IL-13, as measured by flow cytometry and multiplex assays.
  Responders to a specific cytokine were defined as subjects with concentration for that respective cytokine after Bet v 1 stimulation above P95 of the concentration for that cytokine after medium only stimulation for all subjects (Total cohort), AND at least 5 times higher than their own respective concentration after medium only stimulation.
Time Frame: At Day 0
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Allergy Group | Control Group
Number analyzed (Participants) | 10 | 3
Subjects
  IL-13 | 6 | 0
  IL-5 | 7 | 1

3. Secondary Outcome: Number of Subject Responders With Antigen-Th2 CD4+ T Cells Expressing Interferon-gamma (IFN-γ)
Description: Responders are defined as subjects with a concentration after Bet v 1 stimulation above P95 (determined on Bet v 1 BrdU+ subjects) of all concentrations after medium only stimulation
Time Frame: At Day 0
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Allergy Group | Control Group
Number analyzed (Participants) | 10 | 3
Subjects | 8 | 3

4. Secondary Outcome: Number of Subject Responders With Antigen-Th2 CD4+ T Cells Expressing IFN-γ - Amended Definition
Description: Responders to a specific cytokine were defined as subjects with concentration for that respective cytokine after Bet v 1 stimulation above P95 of the concentration for that cytokine after medium only stimulation for all subjects (Total cohort), AND at least 5 times higher than their own respective concentration after medium only stimulation.
Time Frame: At Day 0
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Allergy Group | Control Group
Number analyzed (Participants) | 10 | 3
Subjects | 8 | 2

ADVERSE EVENTS:
Time Frame: SAEs related to study participation/concurrent GSK medication/vaccine reporting was done at Day 0
Arm/Group | Allergy Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.